CLINICAL TRIAL: NCT07230873
Title: The Impact of Stationary Combined Exercise on Adiponectin and High-Sensitivity C-Reactive Protein Levels in Overweight Women
Brief Title: The Impact of Stationary Combined Exercise on Adiponectin and Hs-CRP Levels in Overweight Women
Acronym: SCEX-ADCRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xianjie Zheng (Other)
Responsible Party: Sponsor-Investigator, Xianjie Zheng, College of Physical Education and Health, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: College of Physical Education; K2016038 (Registry Identifier: Ethics Approval Number (Chongqing College of International Business and Economics Research Ethics Committee).)
Record Dates: First submitted 2025-09-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Overweight; Obesity; Inflammation, Low-Grade; Cardiovascular Diseases, Risk Factors
Keywords: Adiponectin; inflammation; combined station training; hs-CRP
MeSH Terms: conditions — Overweight; Obesity; Inflammation; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Exercise Group (Experimental): Arm 1 reflects the circuit-based combined exercise intervention.
  Interventions: Behavioral: Combined Exercise Group
- Control Group (Experimental): Arm 2 reflects the no structured exercise condition.
  Interventions: Behavioral: No Structured Exercise

INTERVENTIONS:
Behavioral: Combined Exercise Group — Participants completed an eight-week circuit-based combined exercise program, four sessions per week, at an intensity of 70-90% of maximum heart rate. Each session began with a 10-15 minute warm-up (stretching and light jogging) and ended with a 5-10 minute cool-down (walking and stretching). The main exercise protocol included six stations (sit-ups, step jumps, push-ups, jump rope, jumping jacks, and medicine ball lifting), performed in three rounds. The duration at each station progressively increased from 60 seconds (weeks 1-2) to 150 seconds (weeks 7-8), with rest intervals of 30-50 seconds between stations and 3-5 minutes between rounds. Exercise intensity was monitored with a Polar heart rate monitor to ensure participants stayed within the target zone.
  Other Names: High-Intensity Circuit-Based Combined Exercise; Combined Stationary Exercise; SCEX Program (Stationary Combined Exercise)
  Arms: Combined Exercise Group
Behavioral: No Structured Exercise — Participants in the control group will not receive any structured exercise program during the eight-week study period. They will be instructed to maintain their usual daily routines and refrain from initiating any new organized exercise or training programs beyond their routine physical education classes and everyday activities.
  Other Names: Usual Activity; No Exercise Program
  Arms: Control Group

SUMMARY:
This study looked at whether a specific exercise program can improve inflammatory markers in overweight young women. We tested an eight-week, circuit-style exercise program that combines aerobic and resistance activities (e.g., sit-ups, step jumps, push-ups, jump rope, jumping jacks, medicine-ball lifts). Participants exercised four times per week at a moderate-to-high intensity, with a warm-up and cool-down at each session.

Twenty-two women (ages 20-30 years; BMI 25-31 kg/m²) were randomly assigned to one of two groups: (1) the exercise group completed the training program; (2) the control group continued usual daily activities without a structured program. Before starting and 48 hours after finishing the program, we took fasting blood samples to measure two markers: adiponectin (a hormone made by fat tissue that supports healthy metabolism and has anti-inflammatory effects) and high-sensitivity C-reactive protein (hs-CRP) (a blood marker of inflammation and cardiovascular risk).

The main outcomes were the changes in adiponectin and hs-CRP from before to after the 8-week period. We also recorded weight, body mass index (BMI), body fat percentage, and fitness (VO₂max). The study was conducted at the Exercise Physiology Laboratory, College of Physical Education and Health, Chongqing College of International Business and Economics (Chongqing, China). The research ethics committee approved the protocol, and all participants provided written informed consent.

Recruitment and data collection are complete. Findings suggest that this circuit-based exercise program can increase adiponectin and lower hs-CRP, alongside improvements in body composition, in overweight young women.

ELIGIBILITY:
Inclusion Criteria:

Female sex Age 20 to 30 years BMI 25 to 31 kg/m² Body weight 63 to 87 kg Generally healthy, without diagnosed chronic illness Willing and able to provide written informed consent Willing to refrain from vigorous physical activity for 48 hours before blood sampling Able to attend 4 supervised training sessions per week for 8 weeks (if assigned to intervention)

Exclusion Criteria:

History of cardiovascular disease, hypertension, or diabetes Current smoking or tobacco use Current use of medications or supplements that affect metabolism or inflammatory markers Pregnancy or breastfeeding Contraindications to moderate-to-high intensity exercise on screening Participation in regular vigorous exercise training within the past 6 months Inability or unwillingness to comply with study procedures (e.g., missing >2 consecutive training sessions)

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Change in Serum Adiponectin Concentration | Baseline and 48 hours post-intervention (end of week 8).
  Serum adiponectin (µg/mL) quantified by ELISA in the fasting state; difference from baseline to 48 hours after completion of the 8-week exercise program.

SECONDARY OUTCOMES:
Change in Serum Adiponectin Concentration | Baseline and 48 hours post-intervention (end of week 8).
  Serum adiponectin (µg/mL) quantified by ELISA in the fasting state; difference from baseline to 48 hours after completion of the 8-week exercise program.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Physical Education and Health, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2024-01-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT07230873/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT07230873/SAP_001.pdf
  • Informed Consent Form (2024-01-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT07230873/ICF_002.pdf